CLINICAL TRIAL: NCT06119191
Title: Clinical Evaluation of Comfilcon A Contact Lenses
Brief Title: Clinical Evaluation of Reusable Soft Contact Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CooperVision International Limited (CVIL) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CV-23-86
Record Dates: First submitted 2023-10-31; First posted 2023-11-07 (Actual); Results first posted 2025-03-26 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-02

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Control Lenses (Experimental): Participants wore Control Lenses for 30±2 days.
  Interventions: Device: Control Lenses (comfilcon A with current process)
- Test Lenses (Experimental): Participants wore Test Lenses for 30±2 days.
  Interventions: Device: Test Lenses (comfilcon A with novel process)

INTERVENTIONS:
Device: Control Lenses (comfilcon A with current process) — Daily wear lenses for 30±2 days
  Arms: Control Lenses
Device: Test Lenses (comfilcon A with novel process) — Daily wear lenses for 30±2 days
  Arms: Test Lenses

SUMMARY:
The purpose of this study was to confirm the clinical performance of a novel manufacturing process for comfilcon A contact lenses in habitual wearers over a one-month period of lens wear.

DETAILED DESCRIPTION:
This was a prospective, multiple day, double-masked (investigator and subject), randomized, bilateral re-fit parallel arm study comparing a Test Lens against an appropriate Control Lens. Participants were randomized to wear the Test or Control lens for 30±2 days.

ELIGIBILITY:
Inclusion Criteria:

* Have had a self-reported oculo-visual examination in the last year.
* Are at least 18 years of age and has full legal capacity to give their informed consent.
* Have read and understood the informed consent letter.
* Are willing and able to follow instructions and maintain the appointment schedule.
* Have a contact lens spherical prescription between -0.50 D to -6.00 D (inclusive)
* Are correctable to a visual acuity of 20/40 or better (in each eye) with their habitual vision correction or 20/20 best-corrected.
* Have spectacle cylinder of ≤ 0.75 D in both eyes.
* Is a habitual comfilcon A wearer and worn a comfilcon A lens for at least one month (minimum of 8 hours a day, 5 days per week)
* Currently employ the use of a peroxide or multipurpose solution cleaning and disinfecting regimen in one of the following brand names:

  * Bausch and Lomb BioTrue Multi-Purpose Solution
  * Bausch and Lomb BioTrue Hydration Plus Multi-Purpose Solution
  * Bausch and Lomb ReNu Advanced Formulation Multi-Purpose Solution
  * Alcon Opti-Free Puremoist with Hydraglyde Multi-Purpose Solution
  * Alcon Opti-Free Replenish Multi-Purpose Solution
  * Alcon Clear Care Plus Hydrogen Peroxide Solution
  * Acuvue RevitaLens Multi-Purpose Solution
* Have clear corneas and no active ocular disease.
* Have not worn habitual lenses for at least 12 hours before the baseline/screening examination
* Are willing to wear the study contact lenses for at least 8 hours per day, 5 days per week

Exclusion Criteria:

* Have never worn contact lenses before.
* Are currently wearing daily disposable contact lenses.
* Have any systemic disease affecting ocular health.
* Are using any systemic or topical medications that will affect ocular health.
* Have any ocular pathology or abnormality that would affect the wearing of contact lenses.
* Have any clinically significant lid or conjunctival abnormalities, active neovascularization or any central corneal scars.
* Are aphakic.
* Have undergone corneal refractive surgery.
* Are participating in any other type of eye related clinical or research study.
* Require a change in lens power from more than 1 diopter as dictated by over-refraction with their habitual lens prescription.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2023-11-14 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Meng C Lin, OD PhD, Principal Investigator — Clinical Research Center, UC Berkeley; Josianne Manasse, OD, Principal Investigator — SUNY College of Optometry Clinical Vision Research Center; Peter Kollbaum, OD PhD, Principal Investigator — Clinical Optics Research Lab at IU School of Optometry; Katherine Bickle, OD, Principal Investigator — ProCare Vision Center, Inc.; Jennifer S Fogt, OD MS, Principal Investigator — Ohio State University
Locations (5):
- United States (5):
  - Clinical Research Center, UC Berkeley, Berkeley, California
  - Clinical Optics Research Lab at IU School of Optometry, Bloomington, Indiana
  - SUNY College of Optometry Clinical Vision Research Center, New York, New York
  - Ohio State University College of Optometry, Columbus, Ohio
  - ProCare Vision Center, Inc., Granville, Ohio

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Three participants did not meet the inclusion criteria and were excluded from the analysis.
Period: Overall Study
Arm/Group | Control Lenses | Test Lenses
Started | 26 | 48
Completed | 25 | 47
Not Completed | 1 | 1
Not completed — Adverse Event | 0 | 1
Not completed — Protocol Violation | 1 | 0

BASELINE CHARACTERISTICS:
Population: All participants that were dispensed intervention (Control or Test Lens) and completed the study
Groups:
- Control Lenses: Participants that received the Control Lens
- Test Lenses: Participants that received the Test Lens
- Total: Total of all reporting groups
Arm/Group | Control Lenses | Test Lenses | Total
Number analyzed (Participants) | 25 | 47 | 72
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.6 (11.0) | 29.0 (8.5) | 29.5 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 29 | 50
  Male | 4 | 18 | 22
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Visual Acuity
Description: Monocular distance logMAR visual acuity at distance 4 meters under high illumination, high contrast conditions was measured at the 4 week timepoint of lens wear.
Time Frame: 4 weeks
Population: Analysis population includes all participants that were eligible (inclusion/exclusion criteria) and completed all study visits.
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Control Lenses | Test Lenses
Number analyzed (Participants) | 25 | 47
logMAR | -0.07 (0.08) | -0.13 (0.08)

ADVERSE EVENTS:
Time Frame: Length of study, approximately 30±2 days
Arm/Group | Control Lenses | Test Lenses
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/48
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/48
Other Adverse Events (participants affected / at risk) | 0/26 | 1/48
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control Lenses (N=26) | Test Lenses (N=48)
Ocular Hyperemia and Discomfort (Eye disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-11-02): https://cdn.clinicaltrials.gov/large-docs/91/NCT06119191/Prot_SAP_000.pdf